CLINICAL TRIAL: NCT01135836
Title: A Randomized, Controlled, Single Blind Study Comparing a Pulmonary Recruitment Maneuver Versus Intraperitoneal Infusion of Normal Saline to Reduce Shoulder Tip Pain After Gynecologic Laparoscopic Surgery
Brief Title: Reducing Shoulder Tip Pain Following Laparoscopic Surgery
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Collaborators: National Yang Ming Chiao Tung University (Other)
Responsible Party: Yi Jen, Chen, M.D., Ph.D., Department of Obstetrics and Gynecology, Taipei Veterans General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: VGHIRB No. 980705
Record Dates: First submitted 2010-06-02; First posted 2010-06-03 (Estimated); Last update posted 2010-06-03 (Estimated); Status verified 2010-06

CONDITIONS: Shoulder Pain; Laparoscopic Surgery
Keywords: Shoulder pain; Gynecologic laparoscopic surgery; Nausea; Vomiting; Abdominal fullness
MeSH Terms: conditions — Shoulder Pain; Nausea; Vomiting | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- pulmonary recruitment maneuver (Experimental): a pulmonary recruitment maneuver consisting of five manual pulmonary inflations was performed with a maximum pressure of 60 cm H2O. The anestheiologist held the fifth positive pressure inflation for approximately 5 seconds.
  Interventions: Procedure: Pulmonary recruitment maneuver
- intraperitoneal normal saline (Experimental): the upper part of the abdominal cavity was evenly and bilaterally filled with the 0.9% normal saline in the amount of 500 cc. We will leave the fluid in the abdominal cavity
  Interventions: Procedure: Intraperitoneal normal saline
- Control group (Placebo Comparator): CO2 was removed by passive exsufflation through the port site.
  Interventions: Procedure: Control group

INTERVENTIONS:
Procedure: Pulmonary recruitment maneuver — a pulmonary recruitment maneuver consisting of five manual pulmonary inflations was performed with a maximum pressure of 60 cm H2O. The anestheiologist held the fifth positive pressure inflation for approximately 5 seconds.
  Arms: pulmonary recruitment maneuver
Procedure: Intraperitoneal normal saline — the upper part of the abdominal cavity was evenly and bilaterally filled with the 0.9% normal saline in the amount of 500 cc. We will leave the fluid in the abdominal cavity.
  Arms: intraperitoneal normal saline
Procedure: Control group — CO2 was removed by passive exsufflation through the port site.
  Arms: Control group

SUMMARY:
Laparoscopic surgery is becoming a major procedure, owing to smaller incisions, shorter hospitalizations, and less post-operative pain as compared with traditional laparotomies. However, there is marked interindividual variability of post-operative shoulder-tip pain following laparoscopic surgery. The incidence of shoulder pain varies from 35% to 80% and ranges from mild to severe. In some cases, it has been reported to last more than 72 hours after surgery.

The hypothesis of post-operative shoulder-tip pain is that carbon dioxide induced phrenic nerve irritation causes referred pain to C4. Therefore, the investigators should try to reduce carbon dioxide retention in the pelvic cavity.

DETAILED DESCRIPTION:
This clinical controlled trial is tried to find out the practical and clinical maneuver to reduce post-operative should-tip pain following laparoscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients receive benign gynaecological laparoscopic surgery.
* American Society of Anesthesiologists (ASA) physical status of patient:

classification I-II

Exclusion Criteria:

* The procedure will be required to conversion to laparotomy.
* Any cardio-vascular diseases.

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2009-08; Primary Completion 2010-09 (Estimated); Study Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
the severity and frequency of shoulder-tip pain after laparoscopic surgery | the first 48 hours after the surgery
  We will follow the patients in the first 48 hours after the surgery. The primary outcome measure of this trial is the severity and frequency of shoulder-tip pain after laparoscopic surgery.
  The main objective of this trial is to assess the efficacy of clinical maneuver to reduce shoulder-tip pain after laparoscopic surgery.

SECONDARY OUTCOMES:
Nausea or abdominal fullness after laparoscopic surgery | the first 48 hours after the surgery
  Postoperative illness, such as nausea, vomiting or abdominal fullness were also recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Jen Chen, Ph.D,, Study Chair — Taipei Veterans General Hospital, Taiwan; Hsiao-Wen Tsai, M.D., Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Tsai HW, Chen YJ, Ho CM, Hseu SS, Chao KC, Tsai SK, Wang PH. Maneuvers to decrease laparoscopy-induced shoulder and upper abdominal pain: a randomized controlled study. Arch Surg. 2011 Dec;146(12):1360-6. doi: 10.1001/archsurg.2011.597. PMID 22184293